CLINICAL TRIAL: NCT01771991
Title: Topical Superoxide Dismutase For the Treatment of Radiation Induced Fibrosis in the Head and Neck Cancer Patient
Brief Title: Study of Topical Superoxide Dismutase to Treat Radiation Induced Fibrosis
Acronym: Sodermix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOD 2012
Record Dates: First submitted 2013-01-11; First posted 2013-01-21 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2017-11

CONDITIONS: Radiation Induced Fibrosis to the Head and Neck
Keywords: fibrosis; radiation; neck; cancer; Sodermix
MeSH Terms: conditions — Fibrosis; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Sodermix Dismutase (Experimental): Patients with measurable radiation induced fibrosis of the neck. Patients will be randomized to applying Topical Sodermix Dismutase in the form of Sodermix(SOD) to the area of neck skin fibrosis twice a day for 12 weeks.
  Interventions: Drug: Topical Sodermix Dismutase in the form of Sodermix (SOD)
- Placebo group (Placebo Comparator): Cetaphil cream
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical Sodermix Dismutase in the form of Sodermix (SOD) — Topical Sodermix Dismutase in the form of Sodermix (SOD) will be applied twice daily, of half dollar application for 12 weeks to fibrosed area.
  Other Names: Sodermix; SOD
  Arms: Topical Sodermix Dismutase
Drug: Placebo — Placebo or cetaphil cream will be applied twice daily, of half dollar size for 12 weeks to fibrosed area.
  Other Names: Cetaphil cream
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine if topical superoxide dismutase is an effective treatment of radiation related neck fibrosis, and to determine the quality of life impact from radiation related fibrosis in the head and neck cancer patients at Sanford Health.

DETAILED DESCRIPTION:
The primary goal of this study is to evaluate the effect of topical Superoxide Dismutase (SOD) on the radiation induced fibrosis in head and neck cancer patients. A prospective, blinded, two group control design will be used with pretest and post test quality of life as well as objective fibrosis assessment. Patients will be randomized to alternatively receive topical SOD or placebo as instructed on twice daily use for 3 months. Pre and post treatment quality of life surveys and objective assessment will determine if the topical SOD improves neck fibrosis/function and global quality of life.

This study will increase clinical trial awareness and participation while potentially improving the long term functional outcomes of head and neck cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* must have evidence of neck fibrosis
* previous radiation treatment to the neck for cancer
* age greater than or equal to 18 years
* life expectancy of greater than 12 weeks
* ability to understand the purpose of the study and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SOD or Cetaphil cram.
* any psychological, familial, sociological or geographical conditions that do not permit medical follow-up and compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C Spanos, MD, Principal Investigator — Sanford Health/Sanford Clinic ENT
Locations (1):
- Sanford Health, Sioux Falls, South Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Sodermix Dismutase: Patients with measurable radiation induced fibrosis of the neck. Patients will be randomized to Topical Sodermix Dismutase in the form of Sodermix(SOD)
  Topical Sodermix Dismutase in the form of Sodermix (SOD): Topical Sodermix Dismutase in the form of Sodermix (SOD) will be applied twice daily, of half dollar application for 12 weeks to fibrosed area.
Period: Overall Study
Arm/Group | Topical Sodermix Dismutase | Placebo Group
Started | 38 | 36
Started Treatment | 37 | 34
Completed | 30 | 30
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Sodermix Dismutase | Placebo Group | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 26 | 54
  >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.98 (9.64) | 61.64 (9.73) | 61.3 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 30 | 29 | 59
Region of Enrollment [Number; unit: participants]
  United States | 38 | 36 | 74

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Neck Fibrosis
Description: Number of participants with improvement in fibrosis as defined as a one point improvement on the fibrosis scale using the grading scale outlined in CTCAE 4.03, page 46.
Time Frame: 3 months
Population: All subjects randomized between August 2012 and May 2013.
Measure: Number; unit: participants
Arm/Group | Topical Sodermix Dismutase | Placebo Group
Number analyzed (Participants) | 38 | 36
participants | 13 | 13

2. Secondary Outcome: Determine the Quality of Life Impact From Radiation Related Fibrosis in Head and Neck Cancer Patients
Description: Metrics are measured via analysis of Health Related Quality of Life questionnaire.
  Functional Assessment of Cancer Therapy for Head and Neck Cancer (FACT H&N) questionnaire was used to evaluate the quality of life in patient receiving treatment of head and neck cancer. Sub-categories of Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, and Head & Neck Additional Concerns are included. Each category used a 5-point Likert scale ranged from 0 to 4 with 0= Not at all (no affect on daily activities) to 4=Very much (significant affect on daily activities).
  Sub-categories were not analyzed individually. All were summed together for total score. Analysis was done comparing baseline scores and end of treatment scores.
  Maximum scale total = 156 (answer of 4 to all items) Minimum scale total = 0 (answer of 0 to all items)
Time Frame: 3 months
Population: The analysis population are those who filled out the Quality of Life questionnaire at baseline and 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical Sodermix Dismutase | Placebo Group
Number analyzed (Participants) | 22 | 20
score on a scale | 2.30 (6.60) | 0.44 (9.17)
Statistical Analysis 1: Comparison: Topical Sodermix Dismutase vs Placebo Group; Test type: Superiority; p = 0.57, Wilcoxon Rank-Sum; sum of scores = 453, Standard Deviation 39.6 — Standard Deviation under the Null hypothesis for each group

3. Secondary Outcome: Determine the Pain From Radiation Related Fibrosis in Head and Neck Cancer Patients
Description: Subjects use the numeric verbal pain rating scale (0-10 scale specified for neck region with "0" being no pain and "10" extreme pain).
  0 - Pain free
  1. - Very minor annoyance-occasional minor twinges
  2. - Minor annoyance-occasional, does not interfere with activities
  3. - Annoying enough to be distracting
  4. - Can be ignored if you are really involved in your work, but still distracting,
  5. - Can't be ignored for more than 30 minutes. Interrupts some activities.
  6. - Can't be ignored for any length of time, but you can still go to work and participate in social activities.
  7. - Make it difficult to concentrate, interferes with sleep, you can still function with effort, prevents doing daily activities
  8. - Physical activity severely limited. You can read and converse with effort. Hard to do anything
  9. - Unable to do anything, Can't bear the pain
  10. - Bad as it could be, nothing else matters
  Differences between baseline scores and 3 month score
Time Frame: From baseline to 3 months.
Population: All patients who had a pre-treatment and post-treatment pain score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical Sodermix Dismutase | Placebo Group
Number analyzed (Participants) | 26 | 30
score on a scale | 0.31 (1.01) | 0.13 (1.81)
Statistical Analysis 1: Comparison: Topical Sodermix Dismutase vs Placebo Group; Looking at the difference in pain change over time. The null hypothesis is there was no difference between the two treatment groups; Test type: Superiority; p = 0.65, t-test, 2 sided; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.60 to 0.95], Standard Deviation 1.50

4. Secondary Outcome: Cervical Spine Range of Motion
Description: Determine the effect of the treatment on Range of Motion over time. Cervical spine rotation was measured by a physical therapist using a goniometer.
  A goniometer is an instrument that either measures an angle or allows an object to be rotated to a precise angular position. Results are documented in degrees.
  Baseline measurements were compared with post-treatment measurements. A larger post-treatment measure when compared to the baseline measurement would indicate an increase of the cervical spine range of motion.
Time Frame: 3 months
Population: Patients with pre-treatment and post-treatment measures.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Topical Sodermix Dismutase | Placebo Group
Number analyzed (Participants) | 29 | 30
degrees | -7.14 (14.27) | -9.77 (20.63)
Statistical Analysis 1: Comparison: Topical Sodermix Dismutase vs Placebo Group; Looking at the difference in range of motion change over time. The null hypothesis is there was no difference between the two treatment groups; Test type: Superiority; p = 0.57, t-test, 2 sided; Mean Difference (Final Values) = 2.63, 95% CI 2-sided [-6.65 to 11.91], Standard Deviation 17.79

ADVERSE EVENTS:
Time Frame: 3 months
Description: During each study visit and telephone interview, scheduled weekly, subjects will be asked open-ended questions to elicit any medically related changes in their well-being.
Arm/Group | Topical Sodermix Dismutase | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/36
Other Adverse Events (participants affected / at risk) | 0/38 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes